CLINICAL TRIAL: NCT04356287
Title: Phase I/II Randomized Controlled Trial of Umbilical Cord-derived mesenChymAl stRomal cElls in Systemic Sclerosis
Brief Title: Treatment With Human Umbilical Cord-derived Mesenchymal Stromal Cells in Systemic Sclerosis
Acronym: CARE-SSc
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Marie Hudson, MD (Other)
Collaborators: Medical University of South Carolina (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Université de Montréal (Other); Assistance Publique - Hôpitaux de Paris (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other); University Paris 7 - Denis Diderot (Other)
Responsible Party: Sponsor-Investigator, Marie Hudson, MD, Rheumatologist, Jewish General Hospital; Physician-scientist, Lady Davis Institute for Medical Research, Sir Mortimer B. Davis - Jewish General Hospital
Organization: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-05-2020-2251
Record Dates: First submitted 2020-04-15; First posted 2020-04-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Sclerosis, Systemic; Mesenchymal Stem Cells
Keywords: Systemic Sclerosis; Umbilical cord-derived mesenchymal stromal cells; Scleroderma, Systemic
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study participants, physicians (including the outcome assessors) and research nurses will be blinded to treatment arm. Only the study statistician and the personnel at the manufacturing laboratory at the Medical University of South Carolina will be aware of the subject's treatment allocation. The Medical University of South Carolina will send blinded infusion bag(s) to the Clinical Research Unit of the Jewish General Hospital.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One infusion of UCMSC (Experimental): Patients receive one intravenous infusion of UCMSC at month 0 and one intravenous infusion of placebo at month 3. Each experimental infusion will consist of 1 million UCMSC/kg suspended in 50 ml of PlasmaLyte A. Each placebo infusion will consist of a similar volume of PlasmaLyte A.
  Interventions: Biological: UCMSC
- Two infusions of UCMSC (Experimental): Patients receive one intravenous infusion of UCMSC at month 0 and one intravenous infusion of UCMSC at month 3. Each experimental infusion will consist of 1 million UCMSC/kg suspended in 50 ml of PlasmaLyte A.
  Interventions: Biological: UCMSC
- Placebo infusions (Placebo Comparator): Patients receive intravenous placebo infusions at months 0 and 3. Each placebo infusion will consist of 50 ml of PlasmaLyte A.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: UCMSC — Each infusion will consist of 1 million MSC/kg suspended in 50 mL of PlasmaLyte A.
  Other Names: umbilical cord derived mesenchymal stromal cells
  Arms: One infusion of UCMSC; Two infusions of UCMSC
Other: Placebo — Each infusion will consist of 50 mL of PlasmaLyte A.
  Arms: Placebo infusions

SUMMARY:
The purpose of this study is to test the safety and efficacy of Umbilical Cord-derived Mesenchymal Stromal Cells (UCMSC) for the treatment of Systemic Sclerosis (SSc).

DETAILED DESCRIPTION:
A single-center, three-arm, randomized, double-blind, placebo-controlled trial is proposed. A total of 18 SSc patients will be enrolled in 3 successive blocks of 6 patients each. After being informed about the study and potential risks, all patients giving written informed consent will be randomized to one of two treatment arms or a placebo arm (total of 6 patients per arm). Within each block, the 6 patients will be randomized in a 2:2:2 ratio in one of the following arms: placebo, 1 infusion of UCMSC (M0), or 2 infusions of UCMSC (M0, M3). Second infusions of UCMSC will be performed only in the absence of Treatment Related Severe Adverse Events (TRSAE). Randomization into blocks 2 and 3 will be staggered, to allow the detection of TRSAE prior to inclusion of patients in a subsequent block, i.e. the second block will be randomized only in the absence of TRSAE one month after the first infusion of all 6 patients in block one, and similarly for the third block.

ELIGIBILITY:
Inclusion Criteria:

1. SSc according to American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) 2103 classification criteria for systemic sclerosis
2. Severe disease defined as:

   i) disease duration of 2 years or less with an mRss of > 20 and (ESR > 25 mm and/or hemoglobin < 11 g/dL, not explained by other causes than SSc), or ii) mRss >15 without any restriction as to disease duration plus at least one major organ involvement as defined by: a) respiratory involvement consisting of lung diffusion capacity for carbon monoxide (DLCO) and/or forced vital capacity (FVC) < 80% predicted and evidence of interstitial lung disease (chest X-ray and/or high resolution computed tomography (HRCT) scan); b) renal involvement consisting of past renal crisis and/or stage 2 or 3 chronic kidney disease (glomerular filtration rate between 30-89 mL/min) not explained by other causes than SSc; c) cardiac involvement consisting of reversible congestive heart failure, atrial or ventricular rhythm disturbances such as recurrent episodes of atrial fibrillation or flutter, recurrent atrial paroxysmal tachycardia, conduction abnormalities (2nd or 3rd degree atrioventricular block), and/or mild to moderate pericardial effusion. All causes of organ involvement should be attributed to SSc.
3. Inadequate response (determined by patient and physician judgement) or adverse events necessitating discontinuation of standard therapy (usually consisting of methotrexate 25 mg subcutaneous (or as tolerated) per week and/or mycophenolate mofetil 2-3 gm/d (or as tolerated) for at least 3 months
4. Ineligibility or unwillingness to undergo autologous hematopoietic stem cell transplant

Exclusion Criteria:

1. Age < 18 years
2. Pregnancy or unwillingness to use adequate contraception
3. Life-threatening end-organ damage defined as:

   * FVC < 45% and/or DLCO (corrected for hemoglobin) < 30% predicted;
   * Left ventricular ejection fraction < 40% by cardiac echocardiography;
   * Pulmonary hypertension with baseline resting systolic pulmonary arterial pressures > 50 mmHg by cardiac echocardiography, or mean pulmonary artery pressure > 25 mmHg (and pulmonary wedge pressure < 15 mmHg) on right heart catheterization;
   * stage 4 or more chronic kidney disease (glomerular filtration rate < 30 ml/min)
4. Liver failure defined as an abnormal transaminase level (aspartate aminotransferase (ASAT), alanine aminotransaminase (ALAT) > 3 normal) unless related to activity of the disease
5. Concurrent neoplasms or myelodysplasia
6. Uncontrolled hypertension
7. Uncontrolled acute or chronic infection (HIV, HTLV-1/2 (Human T-lymphotropic virus), hepatitis B surface Ag positive, hepatitis C positive) or high risk thereof
8. Significant malnutrition with BMI < 18 kg/m2
9. Severe concomitant psychiatric disorder
10. Bone marrow insufficiency defined as neutropenia < 0.5 x 109 cell/L, thrombocytopenia < 30 x 109 cell/L, anemia < 8g/dL, CD4+ T lymphopenia < 200 x 106 cell/L due to other diseases than SSc (CD4 - cluster of differentiation 4)
11. History of poor compliance
12. Concurrent enrolment in any other protocol using an investigational drug
13. Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Measure of safety one month after first infusion | Month 1
  Treatment related severe adverse event using the NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0 classification [https://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm]

SECONDARY OUTCOMES:
Change in modified Rodnan skin score (mRss) between Month 0 and Month 12 | Month 0 and Month 12
  A measure of skin thickness; difference between Month 12 and Month 0 on the mRss [Khanna et al., 2017]

OTHER OUTCOMES:
Safety at the time of infusion, 24 hours, 10 days +/- 24 hours, Month 6, Month 9 and Month 12 (adverse events) | 24 hours, 10 days +/- 24 hours, Month 6, Month 9 and Month 12
  Measure of safety of UCMSC in severe SSc using the NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0 classification [https://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm]
Mortality occurring after randomization and up to study completion | 1 year
  Causes of death and their relation to SSc versus the study intervention will be evaluated by the Data and Safety Monitoring Committee (DSMC).
Modified Rodnan skin score | Month 0, Month 3, Month 6 and Month 9
  A measure of skin thickness [Khanna et al., 2017]
World Health Organization (WHO) performance status | Month 0, Month 3, Month 6, Month 9 and Month 12
  WHO performance status [Oken et al., 1982] describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.).
Scleroderma-Health Assessment Questionnaire | Month 0, Month 3, Month 6, Month 9 and Month 12
  Disease status as measured by the Scleroderma-Health Assessment Questionnaire [Steen & Medsger, 1997]
36-Item Short Form Survey version 2 for health-related quality of life (SF-36v2) | Month 0, Month 3, Month 6, Month 9 and Month 12
  Health-related quality of life as measured by the SF-36v2 [Ware et al., 2007]
EuroQoL health status measure (EQ-5D-5L) | Month 0, Month 3, Month 6, Month 9 and Month 12
  Health related quality of life in cost effectiveness analysis as measured by the EQ-5D-5L [Herdman et al., 2011] using five levels of severity in five dimensions.
Response to treatment | Month 0, Month 12
  Defined as decrease in mRss > 25%, increase in FVC > 10% predicted (forced vital capacity) and/or increase in DLCO >15% predicted (diffusing capacity of the lungs for carbon monoxide), without need for further immunosuppression except low dose steroids
Progression-free survival | Month 0, Month 12
  Progression defined as any one of the following: decrease in FVC > 10% predicted; decrease in DLCO > 15% predicted; decrease in left ventricular ejection fraction on cardiac echocardiography > 15%; decrease in weight > 15%; decrease in creatinine clearance > 30%; increase in mRss > 25%; and/or increase in Scleroderma-Health Assessment Questionnaire > 0.5
Global Rank Composite Score | Month 0, Month 12
  A composite score consisting of a hierarchy of ordered outcomes: death, event-free survival (survival without respiratory, renal, or cardiac failure), FVC, score on the Disability Index of the Health Assessment Questionnaire (HAQ-DI; range, 0 to 3, with higher scores indicating more disability), and the modified Rodnan skin score. [Sullivan et al., 2018]
ACR Provisional Composite Response Index | Month 0, Month 12
  ACR Provisional Composite Response Index for Clinical Trials in Early Diffuse Cutaneous Systemic Sclerosis (CRISS) [Khanna et al., 2016], a composite measure of treatment response in SSc

CONTACTS AND LOCATIONS:
Overall Officials: Marie Hudson, MD, Principal Investigator — Sir Mortimer B. Davis - Jewish General Hospital
Locations (1):
- Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang D, Zhang H, Liang J, Wang H, Hua B, Feng X, Gilkeson GS, Farge D, Shi S, Sun L. A Long-Term Follow-Up Study of Allogeneic Mesenchymal Stem/Stromal Cell Transplantation in Patients with Drug-Resistant Systemic Lupus Erythematosus. Stem Cell Reports. 2018 Mar 13;10(3):933-941. doi: 10.1016/j.stemcr.2018.01.029. Epub 2018 Mar 1. PMID 29478901
- [Background] Liang J, Zhang H, Kong W, Deng W, Wang D, Feng X, Zhao C, Hua B, Wang H, Sun L. Safety analysis in patients with autoimmune disease receiving allogeneic mesenchymal stem cells infusion: a long-term retrospective study. Stem Cell Res Ther. 2018 Nov 14;9(1):312. doi: 10.1186/s13287-018-1053-4. PMID 30428931
- See also: US Department of Health and Human Services. National Cancer Institute Common Terminology Criteria For Adverse Events (CTCAE), Version 5.0. 2017 — https://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm